CLINICAL TRIAL: NCT03703713
Title: Colloid Osmotic Pressure and Osmolality in Hyponatremia. Additional Diagnostic Aspects and Guide to Treatment
Brief Title: Colloid Osmotic Pressure and Osmolality in Hyponatremia
Status: Terminated | Type: Observational
Why Stopped: Changes in hospital routine made enrolement difficult.
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Joachim Zdolsek, MD, PhD, Assoc prof, consultant, University Hospital, Linkoeping
Other Study IDs: COOH
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Hyponatremia
MeSH Terms: conditions — Hyponatremia | interventions — Sodium Chloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyponatremia: Patients treated for hyponatremia (<125 mmol/L Sodium) in the intensive care department.
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Sodium chloride — Treatment with Sodium chloride

SUMMARY:
Hyponatremia (serum sodium of less than 135 mmol/L)is a very common electrolyte disorder. The reasons for the disorder varies as well as if it is acute or chronic.

In this study we wish to follow changes in colloid osmotic pressure and osmolality during the initial treatment hours. We also wish to use mass balance for the calculation of body compartments and to detect fluid translocation between these.

DETAILED DESCRIPTION:
Patients with hyponatremia arriving att the intensive care unit are asked to participate in the study. The first blood samples are collected before initializing the treatment as well as measurements of body compartments with a bioimpedance analyzer. Collected blood samples are electrolytes (Sodium, Potassium and Chloride), colloid osmotic pressure, osmolality and hemoglobin. These samples are repeated at 4 and 8 hours after start of the study. Amount of infused fluid as well as electrolytes are recorded. Urine volume is measured and urine samples are analyzed for the loss of electrolytes.

Additional samples for guidance of treatment are collected every hour.

Hopefully the addition of colloid osmotic pressure, osmolality and mass balance can be beneficial in the diagnosis of the reason for the disorder as well as for the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for Hyponatremia at the intensive care unit.

Exclusion Criteria:

* Circulatory instable patients in need of treatment for more than the hyponatremia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for severe hyponatremia, at the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Colloid osmotic pressure | 8 hours
  Measurement of colloid osmotic pressure

SECONDARY OUTCOMES:
Body compartments | 8 hours.
  Bioimpedance analysis is performed every 4 hours.
Body compartments | 8 hours
  Mass balance Sodium and Chloride

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Unit, Vrinnevi Hospital, Norrköping, Sweden